CLINICAL TRIAL: NCT01445314
Title: Analysis of Stored Data Collected From Individuals Administered Neurobehavioral Assessments on IRB-Approved Protocols
Brief Title: Analysis of Data Collected From Individuals Administered Neurobehavioral Assessments
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070110; 07-C-0110; NCT00459199 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: HIV; Brain Tumors; Neurofibromatosis Type 1
Keywords: Stored Data; Neurobehavioral; Natural History; Behavior; Quality of Life
MeSH Terms: conditions — Brain Neoplasms; Neurofibromatosis 1; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Patients: Infants, children, adolescents, and adults who have taken neurobehavioral assessments as part of a past, current, or future IRB-approved protocol.

SUMMARY:
Background:

* People with chronic illness often are at risk for developing neurobehavioral problems due to effects of the disease or associated treatments. These problems may include cognitive impairments involving problem-solving, remembering things, paying attention, and understanding and using language, or emotional functioning or quality of life.
* The National Cancer Institute Medical Illness Counseling Center Neuropsychology Group has collected data from neurobehavioral evaluations of infants, children, adolescents and adults with chronic illnesses enrolled in NIH protocols since 1987 and continues to collect data from patients enrolled in current protocols.
* The data from these evaluations, along with demographic and medical information are stored in an NIH computer database.
* Investigating the neurobehavioral functioning of patients with chronic illness is important for identifying and monitoring the effects of the disease and treatments over time, determining possible at-risk subgroups, evaluating response to therapy, and recommending educational and rehabilitative interventions.

Objectives:

-To learn about how certain illnesses or treatments may affect a person s cognitive abilities, emotional functioning and quality of life.

Eligibility:

* Patients currently enrolled in NIH studies who are having neuropsychological testing or completing quality-of-life questionnaires as part of that study.
* Data obtained from infants, children, adolescents, and adults administered neurobehavioral assessments as part of a past or future NIH protocol.

Design:

* This study does not involve any extra tests or questionnaires; it uses information collected from evaluations that subjects have already completed or will complete as part of other NIH studies.
* Information about participating patients that may help elucidate how cognitive abilities, emotional functioning, and quality of life are affected in people with chronic illness may be collected and stored.

DETAILED DESCRIPTION:
Background:

Individuals with chronic illness often are at risk for developing neurobehavioral impairments due to effects of the disease and/or associated treatments.

The National Cancer Institute (NCI) Neurobehavioral Group has been collecting neurobehavioral data obtained from the longitudinal psychometric testing of infants, children, adolescents, and adults with various chronic illnesses enrolled on IRB-approved protocols at the NIH since the 1980 s, many of which are now closed. In addition, we continue to collect neurobehavioral data obtained from assessments of individuals enrolled on current IRB-approved protocols.

The neurobehavioral test data from these evaluations, as well as demographic information, medical values, neurologic findings, and neuroimaging abnormalities, are stored in the neuropsychological database currently located on the secure NIH mainframe computer system.

Investigating the neurobehavioral functioning of children with chronic illness is important for identifying and monitoring the effects of the disease and treatments over time, determining possible at-risk subgroups, evaluating response to therapy, and recommending educational and rehabilitative interventions. In addition, the data may be used to compare various aspects of neurobehavioral functioning among different illness groups healthy controls, and validate novel methodologies to better assess selected domains of functioning, such as a pediatric quality of life (QOL) scale for children with chronic illnesses with CNS involvement.

Objective:

To describe the neurobehavioral functioning of individuals with chronic illness based on the analysis of stored data collected from IRB-approved protocols, consisting of retrospective data collected on protocols that are now closed and data collected prospectively on current and future protocols.

Eligibility:

Data obtained from infants, children, adolescents, and adults administered neurobehavioral assessments as part of a past, current, or future IRB-approved protocol.

Design:

No data will be collected specifically for this protocol. Retrospective data previously collected from individuals receiving neurobehavioral assessments as part of past IRB-approved protocols or prospective data that already will be collected as specified in current or future IRB-approved protocols and stored in the secure NCI Neurobehavioral database will be used for data analysis as outlined in this protocol.

Cross-sectional or longitudinal data will be selected from the database for statistical analysis based on the objective being studied. Since different objectives may be studied using various types of data, a variety of statistical analyses will be conducted to examine the stored data depending on the objective being studied.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Data obtained from infants, children, adolescents, and adults administered neurobehavioral assessments as part of a past, current, or future IRB-approved protocol.
  2. Informed consent for subjects greater than or equal to 18 years of age, a legal representative to provide permission for subjects greater than or equal to 18 years who cannot give informed consent, or one parent-legal guardian to provide permission for subjects less than 18 years of age who are administered neurobehavioral assessments after this protocol is approved.
  3. Data obtained from healthy controls, which may be siblings of affected patients, administered neurobehavioral assessments on an IRB-approved protocol.

EXCLUSION CRITERIA:

1. Data may be excluded from a particular analysis if a subject had a CNS condition (i.e., Down s syndrome, severe intraventricular hemorrhage) not related to their primary medical diagnosis (i.e., HIV, cancer) that may affect neurobehavioral functioning, missing values on a particular test being studied, or invalid data as judged by the PI or Chairperson.

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants, children, adolescents, and adults who have taken neurobehavioral assessments as part of a past, current, or future IRB-approved protocol.
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2007-03-23 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Functional | 1 Year
  describe neurobehavioural functioning based on stored data

SECONDARY OUTCOMES:
Validation | 5 years
  validate novel assessment tools
Relationship | 5 years
  relationship between neurobehavioral functioning & medical, neuroimaging, neurologic, and psychiatric variables
Effects | 5 years
  effects of treatment on neurobehavioral functioning over time
Comparison | 5 years
  compare neurobehavioral measures between different subgroups within
Comparison | 5 years
  compare neurobehavioral functioning between different chronic medical conditions
Association | 5 years
  association of neurobehavioral functioning with medication
Adherence & QOL | 5 years
  compare the responses of the patient and caregiver on behavioral adherence & QOL

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Wolters, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Hofman KJ, Harris EL, Bryan RN, Denckla MB. Neurofibromatosis type 1: the cognitive phenotype. J Pediatr. 1994 Apr;124(4):S1-8. doi: 10.1016/s0022-3476(05)83163-4. PMID 8151460
- [Background] Butler RW, Hill JM, Steinherz PG, Meyers PA, Finlay JL. Neuropsychologic effects of cranial irradiation, intrathecal methotrexate, and systemic methotrexate in childhood cancer. J Clin Oncol. 1994 Dec;12(12):2621-9. doi: 10.1200/JCO.1994.12.12.2621. PMID 7989937
- [Background] Tardieu M, Boutet A. HIV-1 and the central nervous system. Curr Top Microbiol Immunol. 2002;265:183-95. doi: 10.1007/978-3-662-09525-6_9. No abstract available. PMID 12014189
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-C-0110.html